CLINICAL TRIAL: NCT03979209
Title: Potential for Cortisol Suppression With the Use of High Volume Nasal Mometasone Irrigations in Varying Dosages.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Advanced Rx (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17121505
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-03

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
Keywords: Cortisol Suppression; Mometasone; Chronic Rhinosinusitis; Steroid Irrigations
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: The sample size is 45 patients. Patients will sign the consent form and get a baseline morning cortisol blood draw to confirm eligibility. Once enrolled, they will be instructed on how to perform the nasal irrigation twice a day with a 240 milliliter saline filled Neilmed bottle. Patients will receive either the 1 milligram mometasone dose, 2 milligram mometasone dose, or 4 milligram of mometasone dose. The dose assignment will be determined by the treating physician. After 12 weeks of continuous use of the mometasone irrigation, there will be a repeat morning blood draw to compare cortisol levels to the baseline blood draw.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mometasone 1mg (Experimental): 1mg capsule dissolved in 240mg saline solution nasal irrigation
  Interventions: Drug: Nasal Mometasone Rinse
- Mometasone 2mg (Experimental): 2mg capsule dissolved in 240mg saline solution nasal irrigation
  Interventions: Drug: Nasal Mometasone Rinse
- Mometasone 4mg (Experimental): 4mg capsule dissolved in 240mg saline solution nasal irrigation
  Interventions: Drug: Nasal Mometasone Rinse

INTERVENTIONS:
Drug: Nasal Mometasone Rinse — Nasal irrigation twice a day (BID) of assigned dose.

SUMMARY:
In the United States, more than 30 million people are diagnosed with sinusitis each year. Moreover, chronic sinusitis effects approximately 15% of the U.S. population and is one of the most common chronic illnesses in America. Budesonide and mometasone nasal sprays are used to relieve sneezing, runny, stuffy, or itchy nose caused by hay fever or other allergies (caused by an allergy to pollen, mold, dust, or pets).

The objective of this study is to determine the incidence of cortisol suppression with the use of mometasone irrigations in varying doses. Low levels of cortisol can cause weakness, fatigue, and low blood pressure.

In using nasal sprays, a drug may enter the body's circulation through direct local absorption in the nasal mucosa or oral absorption of any swallowed medication. Some people can reduce symptom severity using medication, including antihistamines and anti-inflammatory drugs. Nasal irrigation - the flooding of the sinus cavity with warm saline solution - can help to reduce sinus congestion and is often recommended by otolaryngologists for a variety of sinus conditions. The goal of nasal irrigation is to clear excess mucus and foreign debris out of the sinuses, and to moisturize the mucosal membrane. The practice has been subjected to clinical testing and has been found to be safe and beneficial with no apparent side effects.

The addition of budesonide to nasal irrigations has become common practice in the treatment of chronic rhinosinusitis. Mometasone has been shown to be an alternative to budesonide with increased local effects and lower absorption by the body. Studies have shown that saline irrigation treatments show greater effects versus saline spray for providing short-term relief of chronic nasal and sinus symptoms.

There is limited data on the use of mometasone in nasal irrigations. Subjects to be included in the study are those with a diagnosis of chronic rhinosinusitis, with or without nasal polyps and who have had prior endoscopic sinus surgery. This study will test 3 different concentrations of mometasone in a nasal irrigation. Patients will receive either 1 milligram mometasone in their nasal irrigations, 2 milligrams of mometasone, or 4 milligrams of mometasone. The dose assignment will be determined by the treating physician. After 12 weeks of entering this study and use of the mometasone irrigations, there will be a blood draw to compare morning cortisol levels to a baseline blood draw.

DETAILED DESCRIPTION:
Sinusitis is inflammation of the sinuses that results in symptoms such as thickened nasal drainage, nasal congestion and facial pain or pressure. Because sinusitis is often preceded by and almost always accompanied by, inflammation of the nasal mucosa, the term "rhinosinusitis" is used by ENT (ear, nose and throat) physicians to replace the term "sinusitis." Viruses, bacteria, and nasal allergies are common causes of inflammation. The inflamed, swollen mucosa of the nasal and sinus cavities leads to obstruction of the openings of the sinuses. Unable to circulate air and eliminate the secretions that are normally produced, the sinuses then become an ideal environment for bacterial infection.

Sinusitis is categorized into the following types according to the duration of symptoms:

Acute - symptoms are present for 4 weeks or less; Subacute - symptoms are present for more than 4 weeks, but less than 12 weeks; Chronic - symptoms are present for 12 weeks or greater; Recurrent Acute - 4 or more acute episodes occurring within 1 year, with resolution of symptoms between episodes; Acute exacerbation of chronic rhinosinusitis involves an episode of worsening symptoms in a patient with diagnosed with chronic rhinosinusitis.

In the United States, more than 30 million people are diagnosed with sinusitis each year. Moreover, chronic sinusitis effects approximately 15% of the U.S. population and is one of the most common chronic illnesses in America. Both budesonide and mometasone nasal sprays are used to relieve sneezing, runny, stuffy, or itchy nose caused by hay fever or other allergies (caused by an allergy to pollen, mold, dust, or pets). These nasal sprays are in the class of drugs called corticosteroids. They work by blocking the release of certain natural substances that cause allergy symptoms.

The objective of this study is to determine the incidence of cortisol suppression with the use of nasal mometasone irrigations in varying dosages.

Low levels of cortisol can cause weakness, fatigue, and low blood pressure. In using nasal sprays, a drug may enter the body's circulation through direct local absorption in the nasal mucosa or oral absorption of any swallowed medication. Some people can reduce symptom severity using medication, including antihistamines and anti-inflammatory drugs. Nasal irrigation - the flooding of the sinus cavity with warm saline solution - can help to reduce sinus congestion and is often recommended by otolaryngologists for a variety of sinus conditions. The goal of nasal irrigation is to clear excess mucus and foreign debris out of the sinuses, and to moisturize the mucosal membrane. The practice has been subjected to clinical testing and has been found to be safe and beneficial with no apparent side effects.

The addition of budesonide to nasal irrigations has become common practice in the treatment of chronic rhinosinusitis. Mometasone has been shown to be an alternative to budesonide with increased local effects and lower absorption by the body. Studies have shown that saline irrigation treatments show greater effects versus saline spray for providing short-term relief of chronic nasal and sinus symptoms. There is limited data on the use of mometasone in nasal irrigations.

The sample size for this study will be 45 patients. Patients will sign the consent form and get a baseline morning cortisol blood draw to confirm eligibility. Once enrolled, they will be instructed on how to perform the nasal irrigation twice a day with a 240 milliliter saline filled Neilmed bottle. Patients will receive either the 1 milligram mometasone dose, 2 milligram mometasone dose, or 4 milligram of mometasone dose. The dose assignment will be determined by the treating physician. After 12 weeks of continuous use of the mometasone irrigation, there will be a repeat morning blood draw to compare cortisol levels to the baseline blood draw.

Scientific Review:

The addition of budesonide to nasal irrigations has become common practice in the treatment of chronic rhinosinusitis. The dose of budesonide 0.5 milligrams/2 milliliters was chosen as a result of convenience, as budesonide respules are commercially available as an inhalation in the treatment of asthma. Mometasone is an alternative to budesonide with improved pharmacokinetics resulting in increased local efficacy and lower systemic absorption, however, data is limited in its use as a topical irrigation formulation.

There is relevant literature available discussing the pharmacokinetic profile of budesonide and mometasone used intranasally. Following intranasal administration a drug may enter systemic circulation through direct local absorption in the nasal mucosa or oral absorption of any swallowed medication. The intranasal bioavailability of budesonide and mometasone through nasal mucosa have been measured at 34% and less than 0.1% respectively. If a drug enters systemic circulation through the nasal mucosa, the medication is subject to plasma protein binding. When a medication is protein bound it is not bioactive and thus reduces the potential for systemic adverse effects. Approximately 85-90% of budesonide is bound to plasma proteins after entering systemic circulation. Alternatively, mometasone is 99% protein bound at clinically relevant concentrations. Therefore, budesonide is bioactive at 10-15 times the concentration of mometasone in the serum due to plasma protein binding.

A portion of the drug may also be cleared from the sinuses into the throat and swallowed, making it available for gastrointestinal absorption. Medications absorbed through the gastrointestinal tract are subject to first pass hepatic metabolism which largely determines the amount of medication which reaches systemic circulation. Approximately 90% of swallowed budesonide is metabolized by the liver during first pass metabolism7. On the other hand, when mometasone is swallowed and undergoes first pass metabolism, 99% of the drug is eliminated leaving only 1% of the drug to enter the circulation.

A desired pharmacokinetic property of intranasal steroids is high lipophilicity. Higher lipophilicity leads to increased intranasal absorption as well as prolonged retention in the nasal tissue. Longer retention of the steroid in nasal tissue results in increased exposure to the glucocorticoid receptor. The relative lipophilicity of budesonide and mometasone are 3,980 and 50,000 respectively. Thus, mometasone has twelve times higher lipophilicity than budesonide.

There is current relevant data to assess the safety of mometasone administered intranasally. A review of 20 clinical trials with more than 6,000 patients worldwide at doses up to 20 times the recommended daily dose found no detectable effect of mometasone on the hypothalamic-pituitary-adrenal axis (HPA). Additionally, mometasone at high doses, did not cause atrophy to the nasal mucosa. Intranasal mometasone at a dose of 1600 micrograms, which is 4 times the recommended dose administered daily to human volunteers for 29 days showed no incidence of adverse effects. The effects of oral mometasone on HPA axis function has also been studied. Oral mometasone was administered at doses of 2, 4, and 8 milligrams to 24 healthy male volunteers with no significant change in plasma or urinary cortisol from placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Diagnosis of Chronic Rhinosinusitis, with or without nasal polyposis
* History of prior endosopic sinus surgery
* Must include at least ethmoidectomy with maxillary antrostomy

Exclusion Criteria:

* Exposure to systemic corticosteroids within one month of the date of enrolment in to the study.
* Adrenal insufficiency
* Liver disease
* Use of oral estrogens in women
* Morbid obesity (BMI more than 38)
* Concurrent pregnancy
* Use of medications which may alter HPA axis(refer to Drugs that affect HPAA)
* Ciliary dysmotility, cystic fibrosis, sarcoidosis, systemic vasculitis, IgG or IgA deficiency, known pituitary or adrenal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2022-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bobby Tajudeen, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith KA, French G, Mechor B, Rudmik L. Safety of long-term high-volume sinonasal budesonide irrigations for chronic rhinosinusitis. Int Forum Allergy Rhinol. 2016 Mar;6(3):228-32. doi: 10.1002/alr.21700. Epub 2016 Jan 11. PMID 26750509
- [Background] Soudry E, Wang J, Vaezeafshar R, Katznelson L, Hwang PH. Safety analysis of long-term budesonide nasal irrigations in patients with chronic rhinosinusitis post endoscopic sinus surgery. Int Forum Allergy Rhinol. 2016 Jun;6(6):568-72. doi: 10.1002/alr.21724. Epub 2016 Feb 16. PMID 26879335
- [Background] Derendorf H, Meltzer EO. Molecular and clinical pharmacology of intranasal corticosteroids: clinical and therapeutic implications. Allergy. 2008 Oct;63(10):1292-300. doi: 10.1111/j.1398-9995.2008.01750.x. PMID 18782107
- [Background] Sastre J, Mosges R. Local and systemic safety of intranasal corticosteroids. J Investig Allergol Clin Immunol. 2012;22(1):1-12. PMID 22448448
- [Background] Pulmicort(R) [package insert]. Wilmington, DE: AstraZeneca; 2000.
- [Background] Hochhaus G. Pharmacokinetic/pharmacodynamic profile of mometasone furoate nasal spray: potential effects on clinical safety and efficacy. Clin Ther. 2008 Jan;30(1):1-13. doi: 10.1016/j.clinthera.2008.01.005. PMID 18343239
- [Background] Lipworth BJ, Jackson CM. Safety of inhaled and intranasal corticosteroids: lessons for the new millennium. Drug Saf. 2000 Jul;23(1):11-33. doi: 10.2165/00002018-200023010-00002. PMID 10915030
- [Background] Corren J. Intranasal corticosteroids for allergic rhinitis: how do different agents compare? J Allergy Clin Immunol. 1999 Oct;104(4 Pt 1):S144-9. doi: 10.1016/s0091-6749(99)70310-6. PMID 10518811
- [Background] Brattsand, R. What factors determine anti-inflammatory activity and selectivity of inhaled steroids? Eur. Respir. Rev. 1997, 7, 356- 361.
- [Background] Harvey RJ, Debnath N, Srubiski A, Bleier B, Schlosser RJ. Fluid residuals and drug exposure in nasal irrigation. Otolaryngol Head Neck Surg. 2009 Dec;141(6):757-61. doi: 10.1016/j.otohns.2009.09.006. PMID 19932850
- [Background] Nasonex(R) [package insert]. Whitehouse Station, NJ: Merk & CO.,INC; 1997.
- [Background] Davies RJ, Nelson HS. Once-daily mometasone furoate nasal spray: efficacy and safety of a new intranasal glucocorticoid for allergic rhinitis. Clin Ther. 1997 Jan-Feb;19(1):27-38; discussion 2-3. doi: 10.1016/s0149-2918(97)80070-7. PMID 9083706
- [Background] Brannan, M. D., Seiberling, M., Cutler, D. L., Cuss, F. M., & Affrime, M. B. (1996, January). Lack of systemic activity with intranasal mometasone furoate. In JOURNAL OF ALLERGY AND CLINICAL IMMUNOLOGY (Vol. 97, No. 1, pp. 62-62). 11830 WESTLINE INDUSTRIAL DR, ST LOUIS, MO 63146-3318: MOSBY-YEAR BOOK INC.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from patients at Rush UMC who met the criteria for the study from 1/14/2019 to 11/11/2019.
Groups:
- Mometasone 4mg: 4mg capsule dissolved in 240mg saline solution nasal irrigation. Nasal Mometasone Rinse: Nasal irrigation twice a day (BID) of assigned dose.
Period: Overall Study
Arm/Group | Mometasone 1mg | Mometasone 2mg | Mometasone 4mg
Started | 2 | 14 | 0 (No patients were recruited to arm 3 - Mometasone 4mg)
Completed | 2 | 14 | 0 (No patients were recruited to arm 3 - Mometasone 4mg)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: To check the cortisol level suppression after nasal corticosteroid irrigation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mometasone 1mg | Mometasone 2mg | Total
Number analyzed (Participants) | 2 | 14 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 12 | 14
  >=65 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 9 | 10
  Male | 1 | 5 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 1 | 10 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 14 | 16
Diagnosis of Chronic Rhinosinusitis, with or without nasal polyposis [Count of Participants; unit: Participants] | 2 | 14 | 16
History of prior endosopic sinus surgery o Must include at least ethmoidectomy with maxillary antros [Count of Participants; unit: Participants] | 2 | 14 | 16

OUTCOME MEASURES:

1. Primary Outcome: Morning "AM" Serum Cortisol Level
Description: The potential for cortisol suppression will be assessed with "AM" cortisol level after continuous nasal mometasone irrigation.
Time Frame: Morning (AM) at week 12,
Population: The morning "AM" cortisol levels were added for each participant in the arms.
Measure: Median (Full Range); unit: mcg/dL
Arm/Group | Mometasone 1mg | Mometasone 2mg
Number analyzed (Participants) | 2 | 14
mcg/dL | 17.35 [13.1 to 21.6] | 14.48 [9.3 to 24.8]

ADVERSE EVENTS:
Time Frame: 1year 2 months
Description: Morning "AM" serum cortisol levels 12 weeks after treatment.
Arm/Group | Mometasone 1mg | Mometasone 2mg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/14
Other Adverse Events (participants affected / at risk) | 0/2 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/09/NCT03979209/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT03979209/SAP_001.pdf
  • Informed Consent Form (2020-06-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT03979209/ICF_002.pdf